CLINICAL TRIAL: NCT04557163
Title: Drug-drug Interaction Study with TS-142 in Healthy Adult Subjects (concomitant Administration of Itraconazole)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-142-205-01
Record Dates: First submitted 2020-09-18; First posted 2020-09-21 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — TS-142; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects receiving TS-142 and itraconazole (Experimental): Eligible subjects will receive a single dose of 5 mg TS-142 on Day 1. Subjects will also receive twice-a-day of 200 mg itraconazole on Day 3 and an once-daily single dose of 200 mg itraconazole from Day 4 to Day 7 and single dose of 1 mg TS-142 on Day 6.
  Interventions: Drug: TS-142; Drug: Itraconazole

INTERVENTIONS:
Drug: TS-142 — TS-142 will be given as 1 mg per capsule administered orally with water.
Drug: Itraconazole — Itraconazole will given as 50 mg per capsule administered orally with water.

SUMMARY:
This is an open-label, single-center, single-sequence study to evaluate the concomitant effects of the potent CYP3A inhibitor itraconazole on the single-dose pharmakokinetics, safety and tolerability of oral TS-142 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male age 20 to 39 years at the signing of informed consent
* Subjects whose body mass index (BMI) within the range 18.5 - 25.0 kg/m2, exclusive of 25.0
* Subjects who judged by the principal investigator(s) or subinvestigator(s) to be appropriate as a subjects of this study based on the results of screening tests and the tests obtained prior to the administration of the investigational drug. (Those who have no abnormal findings in the physical examination, vital signs, and standard 12-lead ECG in the screening test and the test obtained prior to administration of the investigational drug, and whose clinical test results are within the standard values of the clinical trial site. However, if who showed abnormal findings but not clinically significant, they can be enrolled in clinical trials based on comprehensive consideration of medical viewpoints by the principal investigator(s) or subinvestigator(s).)
* Subjects who understand, and have willingness and ability to read and sign, the informed consent form

Exclusion Criteria:

* Subjects who have any disease and are judged not to be healthy based on the medical viewpoints by the principal investigator(s) or subinvestigator(s)
* Subjects who have an inappropriate history for participation in this study, including hepatic, renal, cardiovascular, hematological, endocrinological, metabolic, respiratory, gastrointestinal, dermatological, neurological, urological, immunological, psychiatric abnormalities or diseases
* Subjects who have any history of drug or food allergies
* Other protocol defined exclusion criteria could apply

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Cmax | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Maximum observed concentration of unchanged form of TS-142 and its metabolite in plasma.

SECONDARY OUTCOMES:
AUC(0-last) | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Area under the concentration-time curve from time zero to time of the last quantifiable concentration of TS-142 and its metabolite in plasma.

OTHER OUTCOMES:
AUC(0-infinity) | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Area under the concentration-time curve from time zero extrapolated to infinite time of TS-142 and its metabolite in plasma.
Tmax | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Time to Cmax of TS-142 and its metabolite in plasma.
T1/2 | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Terminal phase half-life of TS-142 and its metabolite in plasma.
Vz/F | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Apparent Volume of Distribution During Terminal Phase of TS-142 and its metabolite in plasma.
CL/F | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Apparent Oral Clearance of TS-142 and its metabolite in plasma.
λz | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  terminal elimination rate constant of TS-142 and its metabolite in plasma.
AUC(0-24h) | Sampling at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 48 hours post-dose of TS-142 on Day 1 or Day 6, in addition, at 96, 144, 192, 240 hours post-dose of TS-142 on Day 6.
  Area under the concentration-time curve from time zero to time 24 h of TS-142 and its metabolite in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No